CLINICAL TRIAL: NCT00320866
Title: Evaluation of Symptoms, Complications and Side Effects of Adding Medications Continuously To Subcutaneous Infusion (Hypodermoclysis) In Home Care Hospice Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SOR316302CTIL
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2006-05

CONDITIONS: Home Infusion Therapy; Infusion Pumps
Keywords: Hypodermoclysis; Evaluation of Symptoms

INTERVENTIONS:
Device: syringe driver

SUMMARY:
Background: Terminal patients are often unable to swallow and need medications to control symptoms. In these cases medications are administered continuously and subcutaneously by a syringe driver. A syringe driver is an expensive and sophisticated equipment to operate. Hypodermoclysis is a useful and easy alternative used in the homecare setting for hydration.

Objectives:

1. To assess the level of symptoms control by the administration of morphine, metoclopramide and midazolam by hypodermoclysis versus by a syringe driver.
2. To assess the complications and side effects of infusing these medications continuously by hypodermoclysis versus by a syringe driver.

Methods: Patients in the homecare setting who meet the criteria for parentral infusion and suffer: pain, vomit/nausea and/or agitation will be recruited for the study.

A double blind crossover methodology will be used. Each patient will serve as both intervention and control, and both patient and medical staff will be blinded to the medication route administration. A research nurse will administer the medications. Crossover will take place 48 hours thereafter. A research assistant will conduct evaluation of symptoms and side effects for a period of 4 days. A sample size of 27 patients will be included in the study (calculated for a significance level of 95% and power of 80%).

ELIGIBILITY:
Inclusion Criteria:

* Patients in the home care unit that need medication/s continuously subcutaneously with symptoms level of 6 or higher on a visual analogue scale (VAS) for that symptom.

Exclusion Criteria:

1. Patients and caregivers that refuse to participate.
2. Every occasion when the infusion period will be less than 48 hours.
3. Every occasion when the patient and/or main care giver are not able to provide reliable information by the judgment of the medical staff person or research worker.
4. Patients that will need other medications subcutaneously that are not included in the study during their study treatment period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27
Dates: Start 2002-02; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
level of symptoms control

SECONDARY OUTCOMES:
complications and side effects

CONTACTS AND LOCATIONS:
Overall Officials: Sasson Menachem, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Ben-Gurion University of the Negev Sial Research Center for Family Medicine and Primary Care, Beersheba, Israel